CLINICAL TRIAL: NCT07293104
Title: Children in Pancreatic Surgery
Brief Title: Children in Pancreatic Surgery: Indications, Procedures and Outcomes
Acronym: ChiPS
Status: Completed | Type: Observational
Sponsor: Medizinische Hochschule Brandenburg Theodor Fontane (Other)
Responsible Party: Principal Investigator, Richard Hunger, Principal investigator, Medizinische Hochschule Brandenburg Theodor Fontane
Other Study IDs: ChiPS
Record Dates: First submitted 2025-12-05; First posted 2025-12-18 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-10

CONDITIONS: Pancreatic Surgery; Children
Keywords: Chidren; Pancreatic surgery; Surgical outcomes
MeSH Terms: interventions — Pancreaticoduodenectomy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Pancreatic tumor
  Interventions: Procedure: Pancreatoduodenectomy; Procedure: Total pancreatectomy; Procedure: Distal pancreatectomy; Procedure: Anastomosis of the pancreatic duct; Procedure: Incision of the pancreas; Procedure: Internal drainage of the pancreas; Procedure: Local excision destruction pancreas; Procedure: Marsupialization of a pancreatic cyst; Procedure: Segmental pancreatic resection
- Chronic pancreatitis
  Interventions: Procedure: Pancreatoduodenectomy; Procedure: Total pancreatectomy; Procedure: Distal pancreatectomy; Procedure: Anastomosis of the pancreatic duct; Procedure: Incision of the pancreas; Procedure: Internal drainage of the pancreas; Procedure: Local excision destruction pancreas; Procedure: Marsupialization of a pancreatic cyst; Procedure: Segmental pancreatic resection
- Trauma
  Interventions: Procedure: Pancreatoduodenectomy; Procedure: Total pancreatectomy; Procedure: Distal pancreatectomy; Procedure: Anastomosis of the pancreatic duct; Procedure: Incision of the pancreas; Procedure: Internal drainage of the pancreas; Procedure: Local excision destruction pancreas; Procedure: Marsupialization of a pancreatic cyst; Procedure: Segmental pancreatic resection
- Extra-pancreatic neoplasm
  Interventions: Procedure: Pancreatoduodenectomy; Procedure: Total pancreatectomy; Procedure: Distal pancreatectomy; Procedure: Anastomosis of the pancreatic duct; Procedure: Incision of the pancreas; Procedure: Internal drainage of the pancreas; Procedure: Local excision destruction pancreas; Procedure: Marsupialization of a pancreatic cyst; Procedure: Segmental pancreatic resection
- Other diseases
  Interventions: Procedure: Pancreatoduodenectomy; Procedure: Total pancreatectomy; Procedure: Distal pancreatectomy; Procedure: Anastomosis of the pancreatic duct; Procedure: Incision of the pancreas; Procedure: Internal drainage of the pancreas; Procedure: Local excision destruction pancreas; Procedure: Marsupialization of a pancreatic cyst; Procedure: Segmental pancreatic resection

INTERVENTIONS:
Procedure: Pancreatoduodenectomy — Procedure codes: 5-524.1; 5-524.2; 5-524.3
Procedure: Total pancreatectomy — Procedure codes: 5-525.*
Procedure: Distal pancreatectomy — Procedure code: 5-524.0
Procedure: Anastomosis of the pancreatic duct — Procedure codes: 5-527.*
Procedure: Incision of the pancreas — Procedure codes: 5-520.*
Procedure: Internal drainage of the pancreas — Procedure codes: 5-523.*
Procedure: Local excision destruction pancreas — Procedure codes: 5-521.*
Procedure: Marsupialization of a pancreatic cyst — Procedure codes: 5-522.*
Procedure: Segmental pancreatic resection — Procedure codes: 5-524.0*; 5-524-x; 5-524.y

SUMMARY:
Pediatric patients differ in a variety of properties from adult populations, but comprehensive multicenter or population-based data is missing for pancreatic surgery. This study aimed to evaluate indications, complications, and mortality in pediatric pancreatic surgery.

DETAILED DESCRIPTION:
This retrospective observational population-based cohort study analzes the German Diagnostic-Related Group database and included all children with pancreatic procedures between 2010 and 2023. The primary outcomes are mortality rates, complication rates, and sex differences related to surgical indication and pancreatic procedure. Descriptive epidemiological and multivariable regression analyses are performed to identify risk factors of mortality and occurrence of perioperative complications.

ELIGIBILITY:
Inclusion Criteria:

* stationary hospital admission
* pancreatic surgical procedure

Exclusion Criteria:

* unknown sex or age
* admission for pancreas tranplantation

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All persons addmitted to a German hospital between 2010 and 2023. Population-based dataset.
Sampling Method: Non-Probability Sample
Enrollment: 761 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Mortality rate | 30 days
  Perioperative death

SECONDARY OUTCOMES:
Complication rates | 30 days
  Perioperative surgical-related complication

IPD SHARING:
Plan to Share IPD: No
The data is held and provided by the Federal Statistical Office of Germany and the statistical offices of the federal states. Due to data privacy regulations, data sharing is strictly prohibited by German law. Furthermore, the data was evaluated exclusively within the framework of controlled remote data analysis. This meant that we never had direct access to the raw data.